CLINICAL TRIAL: NCT01118819
Title: Phase I Safety Study of Clostridium Novyi-NT Spores in Patients With Treatment-refractory Solid Tumor Malignancies
Brief Title: Safety Study of Clostridium Novyi-NT Spores to Treat Patients With Solid Tumors That Have Not Responded to Standard Therapies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated. An IT injection study of C. novyi-NT in patients with treatment refractory solid tumor malignancies may be viewed at NCT01924689.
Sponsor: BioMed Valley Discoveries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVDCNV1; J08107 (Other: Previous Sponsor)
Record Dates: First submitted 2010-04-13; First posted 2010-05-07 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Solid Tumor Malignancies
Keywords: Phase I; Metastatic Disease; Solid Tumor; Malignancy; Metastases; Clinical trial; Hypoxia; Necrosis
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Hypoxia; Necrosis | interventions — Bacterial Load

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clostridium novyi-NT spores (Experimental)
  Interventions: Biological: Clostridium novyi-NT spores

INTERVENTIONS:
Biological: Clostridium novyi-NT spores — Phase 1 study: It will be an escalating dose design, with no intracohort escalation. The first cohort dose will begin at 1 X 10(5) spores/kg and will escalate by tripling through 5 cohorts up to 100 x 10(5) spores/kg.
  Other Names: bacteria; anaerobic bacteria

SUMMARY:
This protocol will examine the safety of intravenous administration of Clostridium novyi-NT spores in patients with treatment-refractory solid tumor malignancies. This investigational study will measure anti-tumor activity of C. novyi-NT administered intravenously in patients with treatment-refractory solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of an advanced solid tumor malignancy
2. History of prior treatment with at least one line of systemic anticancer therapy, when an approved systemic therapy is available, and no curative option is available for continued treatment.
3. Measurable disease as defined by RECIST 1.1 criteria.
4. At least 4 weeks has elapsed since the completion of major surgery and the patient is fully recovered from this surgery and any post-surgical complications.
5. ECOG performance status of 2 or less.
6. Patient is at least 18 years of age
7. Patient is capable of giving informed consent.
8. Patient of childbearing potential (defined by the clinical sites' standards) is using adequate birth control measures (e.g., barrier method with spermicide; intrauterine device; implantable or injectable hormonal contraceptives; surgical sterilization) for the duration of the study and will continue to use such precautions for 12 months after receiving treatment.
9. Patient has no significant valvular disease (trace or mild valvular stenosis or regurgitation is allowed).
10. Patient is able to stay within 45 minutes driving time of an emergency room for 28 days following discharge.
11. The patient has a caregiver for 28 days after dosing.

Exclusion Criteria:

1. Positive pregnancy test
2. Serum creatinine level > 1.5 x the upper limit of normal (ULN), chronic renal failure requiring hemodialysis or peritoneal dialysis.
3. Patient has any of the following hematologic parameters: Platelet count equal to or less than 100,000/mm3, Hemoglobin less than 9.0 g/dL, or an ANC less than 1,000 /mm3.
4. Oxygen saturation (Sp02) of less than 95% on room air.
5. Mean arterial blood pressure of less than 70 mmHg.
6. Glasgow Coma Score of less than 15.
7. Treatment with an investigational drug within the past 30 days or 5 half-lives of that drug.
8. Documented evidence of primary brain malignancy or brain metastases.
9. Clinically significant ascites or clinical evidence or history of portosystemic hypertension or cirrhosis.
10. Laboratory evidence of hepatic dysfunction indicated by any of the following: bilirubin > 1.5 x the upper limit of normal, AST or ALT above 2.5X the upper limit of normal, alkaline phosphatase above 2.5X the upper limit of normal or an INR greater than 1.3.
11. Patient has a foreign body which in the opinion of the treating investigator could be difficult to manage in case of infection (e.g. prosthetic hip).
12. Clinically significant pleural effusion.
13. Clinically significant pericardial effusion, circumferential pericardial effusion, or any effusion greater than 1.0 cm at any location around the heart.
14. Need for ongoing treatment with an immunosuppressive agent.
15. History of solid organ transplantation (with the exception of a corneal transplant > 3 months prior to screening).
16. History of an ischemic insult in the previous 12 months (myocardial infarction, cerebral vascular accident, ischemic tissue from injury, transient ischemic attack, or clinically significant peripheral vascular disease).
17. Patient has a history of venous stasis resulting in venous stasis ulcers or > 2+ edema.
18. History of a significant medical illness deemed by the principal investigator or local investigators as unsuitable for the trial - for example:

    i. Symptomatic congestive heart failure; ii. Psychiatric Illness/Social Situation that may make study dangerous; and iii. Unstable angina pectoris.
19. Asplenia.
20. Antibiotic allergies which would preclude treatment for a C. novyi-NT infection, in the event that antibiotics are required.
21. Treatment with antibiotics within 2 weeks (14 days) of dosing.
22. Active and clinically significant systemic or localized infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of C. novyi-NT spore administration in patients with advanced solid tumor malignancies will be measured over a 7-day inpatient admission with routine labs and continuous adverse event assessments. | 2 years

SECONDARY OUTCOMES:
Anti-tumor activity of C. novyi-NT spores will be assessed with serial imaging studies such as CT scans and blood-based tumor markers. | 2 years
Pharmacokinetics of the C. novyi-NT spores will be measured in routine blood sampling over the course of the study. | 2 years
The host immune and inflammatory response to C. novyi-NT spores will be measured in routine blood sampling over the course of the study. | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York